CLINICAL TRIAL: NCT05713227
Title: The Effects of Gellan Gum on the Acute Glycaemic and Appetitive Responses to a White Rice Meal and Impact on Energy Intake Over 7 Days
Brief Title: White Rice and Gellan Gum 7 Days Intervention
Acronym: WIGG2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moira Taylor (Other)
Collaborators: University of Copenhagen (Other); Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor-Investigator, Moira Taylor, Associate Professor, University of Nottingham
Organization: University of Nottingham (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 414-1121
Record Dates: First submitted 2022-12-06; First posted 2023-02-06 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: jasmine rice; white rice; gellan gum; glycemic response
MeSH Terms: interventions — gellan gum

STUDY DESIGN:
Intervention Model Description: Randomised crossover placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gellan gum (Active Comparator): White rice test meal boiled in 356 g water containing 5.5g of gellan to each 185g of uncooked rice (50 g of available carbohydrate). Consumed on Day 1 at the study site, then consumed at home once daily for 7 days, then consumed again once at test site at Day 8
  Interventions: Dietary Supplement: Gellan gum
- Control (Placebo Comparator): White rice test meal boiled in 356 g water without gellan gum (50 g of available carbohydrate). Consumed on Day 1 at the study site, then consumed at home once daily for 7 days, then consumed again once at test site at Day 8
  Interventions: Dietary Supplement: White rice

INTERVENTIONS:
Dietary Supplement: White rice — 185 g Jasmine (white) rice boiled in 356 g water
  Arms: Control
Dietary Supplement: Gellan gum — Food grade hydrocolloid polysaccharide 5.5g dissolved in 356g cooking water containing 185g rice
  Arms: Gellan gum

SUMMARY:
Gellan gum (GG) is a food grade polysaccharide produced by fermentation. In-vitro studies and in vivo pilot studies suggest that adding gellan gum to rice during cooking might reduce the extent of the increase in circulating blood glucose seen after its consumption (glycaemic response). This study will explore whether such a modification in response is sustained, particularly over a period of 7 days of consumption.

DETAILED DESCRIPTION:
BACKGROUND: Rice is a carbohydrate-rich staple source of food for around half of the world population. Consumption is estimated to be 480 million tonnes per year. According to The Food and Agriculture Organization of the United Nations (FAO), rice is easily accessible to people in Asia, Pacific region, parts of Latin America and the Caribbean and, increasingly in Africa. Rice plays an important role in achieving an adequate dietary intake in these countries.

However high consumption of white rice has been linked with high obesity rates and increased risk for type 2 diabetes . However, it is still the favoured type of rice among consumers, contributing to the observed increasing trends in diet-related diseases in countries with high rice consumption . Modifying the properties of white rice products (e.g. reducing the glycaemic index and/or increasing satiety) with relatively simple interventions can contribute to producing foods that may promote better health due to modified digestion and post prandial metabolic and appetitive profiles. One way to reduce the glycaemic index of white rice may be the addition of hydrocolloids. These have previously been shown to modify the digestibility of foods . The health advantage derived from such modifications would be beneficial for consumers worldwide. Preliminary in-house in vitro digestion data suggested that the addition of gellan gum to rice cooking may reduce digestibility rates though mechanisms yet to be understood. Gellan gum (GG) "is a high molecular weight, water-soluble anionic, extracellular polysaccharide which is produced by the microorganism Sphingomonas elodea during fermentation". GG is commonly used as a gelling agent in foods. Gels formed by gellan gum have high resistance to acid, heat, and enzyme activity. The United States Food and Drug Administration (FDA) has approved the use of GG as a food additive for the human consumption (US.FDA, 2018). It is also approved by the European Community as a food additive with code (E-418). Gellan Gum is gluten free and broadly applied in gluten free foods to provide improved texture and good taste to pasta, biscuits, candy and dairy products. Therefore, it has been proved safe in the amounts the investigators intend to use, it is also suitable for people diagnosed with Coeliac disease as well as suitable for vegetarians, kosher and Halal diets, which make it acceptable for consumption and dietary intervention across different populations.

AIM: The overall purpose of this study is to explore the impact of cooking rice with gellan on the glycaemic and appetitive responses in healthy participants. Both the acute response to one meal will be considered, and the impact on the acute response having consumed the rice once a day over the preceding 7 days. Tolerance will also be considered.

HYPOTHESIS: This work will test the hypothesis that the addition of gellan gum to jasmine rice during cooking will reduce the post prandial glycaemic response. The investigators will also explore associated food intake, appetitive responses and tolerance during both the acute single meal exposure and over a 7 day period of consuming the same portion of rice each day, therefore testing the stability of the glycaemic and appetitive responses after a 7 day period of consumption. Establishing that any acute effect noted is sustained over a period of consumption will be important prior to recommending the addition of gellan to rice cooking as a therapeutic or public health strategy.

ELIGIBILITY:
Inclusion Criteria:

* Not currently taking any medications (except the oral contraceptive pill)
* Aged 18-65 years old
* Body mass index (BMI) ≥ 18.5 and ≤ 24.9 kg/m2
* Able to give informed consent
* Apparently healthy: no medical conditions or previous gastrointestinal surgery which might affect study measurements.

Exclusion Criteria:

* Fasting finger prick screening blood sugar level higher than 5.4 mmol/L
* Restrained eating behaviour as determined by Eating habits and SCOFF screening questionnaires
* Participation in another nutritional or biomedical trial 3 months before the pre-study screening or during the study.
* Reported participation in night shift work during the two weeks prior to pre-study investigation or during the study. Night work is defined as working between midnight and 6.00 AM.
* Strenuous exercise for more than 10 hours per week.
* Consumption of ≥21 alcoholic drinks in a typical week
* Reported weight loss or gain ≥ 10 % of bodyweight during the six months period before the pre-study examination.
* Following a medically- or self-prescribed diet during the two weeks prior to the pre-study examination and until the end of the study
* Dislike of the products served as the dietary test treatments
* Any allergy or food intolerance to the test treatments
* Pregnancy or breastfeeding declared by candidate
* Antibiotic or prescribed probiotic treatment in the past 12 weeks
* Poor understanding of the spoken and/or written English language
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Profile of post prandial 2 hour circulating blood glucose curve | Over 2 hours post consumption
  Fingerprick blood glucose profile for 2 hours post consumption of test rice samples.

SECONDARY OUTCOMES:
Profile of post prandial 3.5 hour circulating blood glucose curve | Over 3.5 hours post consumption
  Fingerprick blood glucose profile for 3.5 hours post consumption of test rice samples rs
Time to Peak of blood glucose | Time period (during the 3.5 hour study period) until peak occurs in hours
  Fingerprick blood glucose time to peak
Peak blood glucose | During the 3.5 hour period of the study.
  Fingerprick blood glucose peak value
Appetite scores post prandial up to 3.5 hours up to 3.5 hours | Over 3.5 hours
  Curve of Visual Analogue Scores up to 3.5 hours postprandially
Gastrointestinal tolerance scores up to 3.5 hours | Over 3.5 hours
  Symptom scores up to 3.5 hours postprandially
Total amount of energy consumed on the first day | Over 24 hours
  Food intake measured from food diaries
Explorative correlations | Over 2 hours and over 3.5 hours
  Explorative correlations between Fingerprick blood glucose area under the curve for 2 hours and 3.5 hours and respectively Area under the curve of appetite Visual Analogue Scores up to 2 hours and 3.5 hours postprandially
Daily appetite scores measured using visual analogue scales | Daily for 7 days
  Appetite score recorded twice daily morning and evening for 7 days using 100mm visual analogue scales with a minimum value of 0mm and maximum value of 100mm.
Gastrointestinal tolerance visual analogue scores questionnaire | Daily for 7 days
  Symptom scores measured daily over 7 days using 100mm visual analogue scales with 0mm as as the minimum and 100mm as the maximum.
Gastrointestinal tolerance categorical questionnaire | Daily for 7 days
  Symptom scores measured daily over 7 days using categorial scores with 0 as as the minimum and 3 as the maximum.
Daily total amount of energy consumed | Daily for 7 days
  Food intake measured from food diaries daily for 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Moira A Taylor, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be available after publication
Supporting Information: Study Protocol, SAP
Time Frame: After publication
Access Criteria: Access on demand

REFERENCES:
- [Background] Garcia MC, Alfaro MC, Calero N, Munoz J. Influence of polysaccharides on the rheology and stabilization of alpha-pinene emulsions. Carbohydr Polym. 2014 May 25;105:177-83. doi: 10.1016/j.carbpol.2014.01.055. Epub 2014 Jan 27. PMID 24708967
- [Background] Azadbakht L, Haghighatdoost F, Esmaillzadeh A. White Rice Consumption, Body Mass Index, and Waist Circumference among Iranian Female Adolescents. J Am Coll Nutr. 2016 Aug;35(6):491-499. doi: 10.1080/07315724.2015.1113902. Epub 2016 Jun 17. PMID 27314887
- [Background] Golozar A, Khalili D, Etemadi A, Poustchi H, Fazeltabar A, Hosseini F, Kamangar F, Khoshnia M, Islami F, Hadaegh F, Brennan P, Boffetta P, Abnet CC, Dawsey SM, Azizi F, Malekzadeh R, Danaei G. White rice intake and incidence of type-2 diabetes: analysis of two prospective cohort studies from Iran. BMC Public Health. 2017 Jan 31;17(1):133. doi: 10.1186/s12889-016-3999-4. PMID 28137245
- [Background] Mond JM, Myers TC, Crosby RD, Hay PJ, Rodgers B, Morgan JF, Lacey JH, Mitchell JE. Screening for eating disorders in primary care: EDE-Q versus SCOFF. Behav Res Ther. 2008 May;46(5):612-22. doi: 10.1016/j.brat.2008.02.003. Epub 2008 Feb 14. PMID 18359005
- [Background] Yi Y, Jeon HJ, Yoon S, Lee SM. Hydrocolloids Decrease the Digestibility of Corn Starch, Soy Protein, and Skim Milk and the Antioxidant Capacity of Grape Juice. Prev Nutr Food Sci. 2015 Dec;20(4):276-83. doi: 10.3746/pnf.2015.20.4.276. Epub 2015 Dec 31. PMID 26770915